CLINICAL TRIAL: NCT06092424
Title: Comparative Study of Pulmonary Artery Pressure (PAP) and Other Hemodynamics Assessed by Echocardiography in Patients With Pulmonary Vascular Diseases Permanently Residing Above 2500 Meters When Assessed Near Resident High Altitude (HA) at 2840m vs. at Low Altitude (LA) Sea Level
Brief Title: High Altitude (HA) Residents With Pulmonary Vascular Diseseases (PVD), Pulmonary Artery Pressure (PAP) Assessed at HA (2840m) vs Sea Level (LA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PVD_HAvsLA_PAP
Record Dates: First submitted 2023-08-09; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Vascular Disease; Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension
Keywords: pulmonary hypertension; Pulmonary Vascular Disease; Chronic Thromboembolic Pulmonary Hypertension; high altitude; hypoxia; pulmonary artery pressure; arterial blood gases
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Altitude Sickness; Hypoxia

STUDY DESIGN:
Intervention Model Description: Patients will be investigated at high altitude (HA, 2840m) and low altitude (LA, sea level)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigations at High altitude (HA, 2840m) (Active Comparator): PAP and other hemodynamics assessed by echocardiography and blood gases near their living altitude in Quito at 2840m
  Interventions: Behavioral: Relocation from HA to LA
- Investigations at Low altitude (LA, sea level) (Experimental): PAP and other hemodynamics assessed by echocardiography and blood gases after the first and second night at LA (sea level)
  Interventions: Behavioral: Relocation from HA to LA

INTERVENTIONS:
Behavioral: Relocation from HA to LA — Patients will be relocated by bus from Quito (2840m) to Pedernales (sea level) and have investigations at both altitudes

SUMMARY:
To study the effect of relocation from 2840m (Quito) to sea level (Pedernales) in patients with pulmonary vascular diseases (PVD) defined as pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension (PH) who permanently live >2500m on pulmonary artery pressure (PAP) and other hemodynamics.

DETAILED DESCRIPTION:
This research in patients with PVD diagnosed with precapillary PH with right heart catheterization and classified to groups 1 and 4 (PAH or CTEPH) who permanently live at HA >2500 (PVD_HA) will have PAP and other hemodynamics assessed by echocardiography and blood gases near their living altitude in Quito at 2840m and at sea level in Pedernales the day after the first and the second night after relocation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-90 years old of both genders,
* Residence > 2500m of altitude
* diagnosed with precapillary PH (mean pulmonary artery pressure (mPAP) >20 mmHg, pulmonary artery wedge pressure (PAWP) ≤15 mmHg and pulmonary vascular resistance (PVR) ≥2 wood units (WU) by right heart catheterization) with PH being classified as PAH or CTEPH according to guidelines
* Patients stable on therapy
* New York Heart Association (NYHA) functional class I-III
* Provided written informed consent to participate in the study.

Exclusion Criteria:

* Age <18 years or >80 years
* unstable condition
* Patients who cannot follow the study investigations, patient permanently living < 2500m.
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, severe smokers (>20 cigarettes/day)
* Severely hypoxemic patients at Quito permanently have persistent oxygen saturation by pulse-oximetry (SpO2) <80% on ambient air.
* Patients with chronic mountain sickness (Hemoglobin > 19 g/dl in women, >21 g/dl in men)
* Patient with a non-corrected ventricular septum defect
* Relevant concomitant other disease of the heart, kidney, liver, blood (anemia hemoglobin<11 g/dl)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary artery Pressure (PAP) in the morning of second day at sea level (LA) | in the morning of the second day at sea level
  Change in PAP in mmHg assessed by echocardiography between LA (sea level) vs High altitude (HA)

SECONDARY OUTCOMES:
Cardiac output in the morning of the second day at sea level | in the morning of the second day at sea level
  Change in cardiac output in l/min assessed by echocardiography between LA (sea level) vs HA (2840 m)
Cardiac output in the morning of the third day at sea level | in the morning of the third day at sea level
  Change in cardiac output in l/min assessed by echocardiography between LA (sea level) vs HA (2840m)
Tricuspid pressure gradient by echocardiography in the morning of the second day at sea level | in the morning of the second day at sea level
  Tricuspid pressure gradient assessed by echocardiography between LA (sea level) vs HA (2840m)
Tricuspid pressure gradient by echocardiography in the morning of the third day at sea level | in the morning of the third day at sea level
  Tricuspid pressure gradient assessed by echocardiography assessed by between LA (sea level) vs HA (2840m)
Tricupsid annular plane systolic excursion by echocardiography in the morning of the second day at sea level | in the morning of the third day at sea level
  Tricupsid annular plane systolic excursion assessed by echocardiography assessed by between LA (sea level) vs HA (2840m)
Tricupsid annular plane systolic excursion by echocardiography in the morning of the third day at sea level | in the morning of the third day at sea level
  Tricupsid annular plane systolic excursion by echocardiography assessed by between LA (sea level) vs HA (2840m)
ph by arterial blood gases in the morning of the second day at sea level | in the morning of the second day at sea level
  Change in ph by arterial blood gases assessed between LA (sea level) vs HA (2840m)
partial pressure of oxygen (PaO2) by arterial blood gases in the morning of the second day at sea level | in the morning of the second day at sea level
  Change in partial pressure of oxygen (PaO2) assessed by arterial blood gases between LA (sea level) vs HA (2840m)
partial pressure of carbon dioxide (PaCO2) by arterial blood gases in the morning of the second day at sea level | in the morning of the second day at sea level
  Change in partial pressure of carbon dioxide (PaCO2) assessed by arterial blood gases partial pressure of carbon dioxide (PaCO2) between LA (sea level) vs HA (2840m)

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Upon request to the PI and after publication of results, data will be shared upon reasonable research questions and ethical approval